CLINICAL TRIAL: NCT03494673
Title: Research of Brain White Matter Hyperintensity in Migraine Using a Cerebrovascular Reactivity Mapping Based on BOLD MRI
Brief Title: Prediction of WMH in Migraine Using a BOLD-CVR Map
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Chin-Sang Chung, MD, PhD, Professor of neurology, Samsung Medical Center
Other Study IDs: 2017-04-049
Record Dates: First submitted 2018-03-28; First posted 2018-04-11 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Migraine
Keywords: White matter hyperintensity; Cerebrovascular reactivity
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Normal controls without headaches will undergo BOLD MRI with prospective CO2 targeting
  Interventions: Diagnostic Test: BOLD MRI
- Migraineurs: Patients diagnosed with migraine based on the ICHD-3 beta will undergo BOLD MRI with prospective CO2 targeting
  Interventions: Diagnostic Test: BOLD MRI

INTERVENTIONS:
Diagnostic Test: BOLD MRI — 1. Prospective End-tidal targeting RespirAct device(A specially designed gas blender and sequential rebreathing circuit) will be used to implement the gas targeting method which involves precise elevations in End-tidal PCO2 while maintaining a fixed End-tidal PO2
  2. BOLD MR images will be obtained by using a T2*-weighted two-dimensional gradient-echo sequence with echoplanar readout.

SUMMARY:
Brain white matter hyperintensities (WMHs) are prevalent in migraineurs, of which the mechanism is still unclear. The investigators aimed to test the spatial association between areas with reduced cerebrovascular reactivity (CVR) to hypercapnic stimuli and consequent development of WMHs.

DETAILED DESCRIPTION:
A whole-brain map of CVR will be created in patients with migraine and normal controls. Hypercapnic stimuli for CVR will be delivered by prospective end-tidal CO2 targeting device. Hemodynamic responses will be determined by BOLD signal changes using fMRI. WMHs will be determined by high-resolution 3D FLAIR imaging. Patients and controls will undergo serial MRIs with 1 year interval. Associations between areas of reduced CVR and consequent WMH development will be tested in both patients and controls.

ELIGIBILITY:
Inclusion Criteria:

1. Migraineurs(patients) :

   * age 18-50 years
   * migraine with or without aura as defined by the third edition of the International Classification of Headache Disorders (ICHD-3 beta)
   * migraine duration > 6 months
   * episodic migraine feature headache (< 15 attacks/m)
   * not any preventive medications for migraine
2. Control:

   * age 18-50 years
   * no headache disorder requiring painkillers within the past year
   * no more than moderate intensity of headache within the past year
   * no headache disorder other than Infrequent episodic tension-type headache as defined by the ICHD-3 beta

Exclusion criteria:

* chronic migraine within last month (≥15 attacks/m)
* medication overuse headache as defined by ICHD-3 beta
* other comorbid disease that may affect vascular function (Hypertension, diabetes, hyperlipidemia, cerebral infarction, smoking etc)
* can not breath 20 L for 1 minute because of basal cardiopulmonary disease (chronic obstructive pulmonary disease, heart failure etc)
* a disease that can be exacerbated by elevated PCO2 in blood (Interstitial lung disease, amyotrophic lateral sclerosis etc)
* predicted to be unable to write the headache diary due to cognitive decline
* contraindications to MRI
* pregnancy
* refusal to informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Controls and migraineurs who visited to a single university hospital
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
CVR association with WMH development | 1-year follow-up (2nd year)
  The investigators will obtain a CVR map using BOLD MR signal in the first year of study and also obtain changes in WMH during 2 years of follow-up period in patients and controls, respectively. Then the investigators will test whether CVR-map predicts consequent WMH development in patients and controls, respectively.

SECONDARY OUTCOMES:
Spatial pattern of CVR | baseline(1st year)
  The investigators will obtain a CVR map for each voxel using BOLD MR signal in response to % increase in EtCO2 respectively in patients and controls. Spatial pattern of CVR will be compared between patients and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Mi Ji Lee, MD, Study Director — Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Seoul, South Korea